CLINICAL TRIAL: NCT05131373
Title: A Phase I, Multi-center, Double-blind, Randomized, Dose Escalating, Parallel Group, Placebo-controlled Safety, Tolerability and Immunogenicity Study of ORI-A-ce001 for the Treatment of Facial Acne Vulgaris
Brief Title: Safety, Tolerability, and Immunogenicity of ORI-A-ce001 for the Treatment of Acne Vulgaris
Acronym: OREA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORI-101-PAC; VBE00004 (Other: Sanofi Identifier); U1111-1294-8125 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-10-11; First posted 2021-11-23 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Acne Vulgaris; Acne
Keywords: acne vulgaris; C. acnes; vaccine; dose escalation; first in human; FIH; skin microbiome; placebo
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1 (Experimental): C. acnes vaccine in adjuvanted formulation will be administered in double-blind fashion in 3 single increasing doses given i.m.
  Interventions: Drug: ORG101 - Experimental 1
- Placebo 1 (Placebo Comparator): Placebo in adjuvanted formulation will be administered in double-blind fashion in single i.m. injections
  Interventions: Drug: ORG101PL - Placebo 1

INTERVENTIONS:
Drug: ORG101 - Experimental 1 — C. acnes vaccine Injection, 25 mcg, 75 mcg, 225 mcg, 4 single i.m. injections given in monthly intervals
  Arms: Experimental 1
Drug: ORG101PL - Placebo 1 — Injection, sterile aqueous solution of aluminium hydroxide, 4 single i.m. injections given in monthly intervals
  Arms: Placebo 1

SUMMARY:
Acne vulgaris, or acne, is one of the most prevalent diseases worldwide, with skin conditions being one of the top causes of years lived with disability and non-fatal disease burden. Despite being one of the most prevalent diseases worldwide, the most widely used treatments in acne have changed little in the past 30 years. To date there is still no effective treatment that can prevent and cure this disease. The currently available acne therapies have been discovered several decades ago, and almost no progress was made in developments of novel, breakthrough treatment approaches.

The present randomized, placebo-controlled, dose escalation, Phase 1 trial (ORI-101-PAC) is intended to investigate the safety, tolerability and immunogenicity of an acne vulgaris vaccine (ORI-A-ce001) at three different dose levels in subjects aged ≥18 years suffering from moderate facial acne vulgaris who are otherwise healthy. The present study will also generate preliminary data on efficacy (inflammatory and non-inflammatory acne lesion counts, acne severity), immunogenicity and functionality of the vaccine, as well as a possible impact on skin microbiome composition. Control groups receiving placebo are included. Data from this trial will be used to inform the design of future studies.

ELIGIBILITY:
Inclusion Criteria: - Male or female subject aged ≥18 years at the time of informed consent signature

* Female subjects of childbearing potential must have a negative serum or urine pregnancy test at Screening and before vaccination and must be willing to practice a highly effective method of contraception during the study
* Subject with a clinical diagnosis of moderate facial acne vulgaris (grade 3 on a 5-grade IGA scale) at Baseline Visit
* Subject must have a maximum of 40 non-inflammatory acne lesions (open and closed comedones) and between a minimum of 20 and a maximum of 70 inflammatory acne lesions (papules and pustules) and a maximum of 1 nodulocystic lesion (nodules and cysts) on the face (e.g., forehead, nose, cheeks, chin, upper lip) at Baseline Visit
* Negative Covid test at Baseline Visit Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Subject who is pregnant, lactating or is planning a pregnancy during the study period
* Subject who has active nodulocystic acne, acne conglobata, acne fulminans, secondary acne or other forms of acne
* Subject who has more than one facial nodules/cysts (where nodule/cyst is defined as an inflammatory lesion greater than or equal to 0.5 cm in size with or without cystic changes)
* Subject who has any skin pathology or condition that, in the Investigator's opinion, could interfere with the evaluation of the Investigational Medicinal Product (IMP) or requires use of interfering topical, systemic, or surgical therapy
* Subject with excessive facial hair, facial skin disorders, skin reactions that may interfere with the study assessments in the Investigator's opinion or skin infection
* History of Guillain-Barré-Syndrome
* Subject who has used any acne-affecting treatment without an appropriate washout period
* Subject who receives active or passive vaccination within 30 days prior to Baseline - Visit Initiation or change of hormonal contraceptive use within 12 weeks prior to Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited and unsolicited local and/or systemic adverse events (AEs) | 7 days following each vaccination
  Number of participants with AEs as assessed by electronic diary (eDiary) and/or PI assessment, and compared to placebo
Incidence of AEs and serious adverse events (SAEs) | Through study completion, an average of 9 months
  Incidence of AEs and SAEs
Number of participants with AEs or SAEs as assessed by physical examination | Through study completion, an average of 9 months
  Number of participants with AEs or SAEs as assessed by physical examination, vital signs, local skin responses, as assessed by treatment arm (vaccine and placebo)
Change from the baseline in laboratory data | Through study completion, an average of 9 months
  Clinically significant change from the baseline in laboratory data as compared to placebo
Change from the baseline in vital signs | Through study completion, an average of 9 months
  Clinically significant change from the baseline in vital signs as compared to placebo
Change from the baseline in ECG | Weeks 0 and 36
  Clinically significant change from the baseline in electrocardiogram (ECG) as compared to placebo
Change from the baseline in physical examination | Through study completion, an average of 9 months
  Clinically significant change from the baseline in physical examination, as compared to placebo

SECONDARY OUTCOMES:
Immunogenicity assessment | Weeks 0, 4, 8, 12, 16, 24 and 36
  The amount of vaccine-antigen-specific serum antibody titers (IgG), measured by ELISA, compared to placebo and compared among different treatment groups
Change in inflammatory lesion counts | Weeks 4, 8, 12, 16, 20, 24, 28, 32 and 36
  Absolute and percentage change from Baseline in the number of inflammatory acne lesions
Change in non-inflammatory lesion counts | Weeks 4, 8, 12, 16, 20, 24, 28, 32 and 36
  Absolute and percentage change from Baseline in the number of non-inflammatory acne lesions
Investigator's global assessment (IGA) - change from Baseline | Weeks 4, 8, 12, 16, 20, 24, 28, 32 and 36
  Absolute change in IGA score from Baseline [scores: 0-4; 0=clear, 4=severe]
Investigator's global assessment (IGA) - percentage of subjects with improvement | Weeks 4, 8, 12, 16, 20, 24, 28, 32 and 36
  Percentage of subjects with at least one-grade improvement in their Baseline IGA score (assessment of mild, clear or almost clear) [scores: 0-4; 0=clear, 4=severe]
Assessment of subjects' treatment acceptability | Week 16
  Treatment acceptability, as assessed by the pre-defined questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Germany (6):
  - Universitäts-Hautklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, North Rhine-Westphalia
  - Universitaetsklinikum der Ruhr-Universitaet Bochum (UKRUB), Bochum, North Rhine-Westphalia
  - CentroDerm, Wuppertal, North Rhine-Westphalia
  - UKSH, Campus Lübeck, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org